CLINICAL TRIAL: NCT02848001
Title: A Phase 1, Open-label, Dose Finding Study of CC-90009, a Novel Cereblon E3 Ligase Modulating Drug, in Subjects With Relapsed or Refractory Acute Myeloid Leukemia or Relapsed or Refractory Higher-Risk Myelodysplastic Syndromes
Brief Title: A Dose-finding Study of CC-90009 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia or Relapsed or Refractory Higher-risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial terminated because of lack of efficacy in the short term acute phase.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90009-AML-001; 2017-001535-39 (EudraCT Number)
Record Dates: First submitted 2016-06-22; First posted 2016-07-28 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: CC-90009; Hematologic Cancers; Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — CC-90009

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC-90009 - Part A (Experimental): Will be administered intravenously per dosing schedule in a 28-day cycle.
  Interventions: Drug: CC-90009
- CC-90009 - Part B - AML and MDS patients (Experimental): Relapsed or refractory AML and MDS subjects. IP will be administered intravenously per dosing schedule determined in Part A
  Interventions: Drug: CC-90009

INTERVENTIONS:
Drug: CC-90009 — CC-90009

SUMMARY:
CC-90009-AML-001 is a phase 1, open-label, dose escalation and expansion, study in subjects with relapsed or refractory acute myeloid leukemia and relapsed or refractory higher-risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
Study CC-90009-AML-001 is an open-label, Phase 1, dose escalation and expansion, first-in-human clinical study of CC-90009 in subjects with relapsed or refractory acute myeloid leukemia (AML) and relapsed or refractory higher-risk myelodysplastic syndrome.

The dose escalation part (Part A) of the study will evaluate the safety and tolerability of escalating doses of CC-90009 in relapsed and refractory AML. The expansion part, (Part B), will further evaluate the safety and efficacy of CC-90009 administered at or below the maximum tolerated dose (MTD) in selected expansion cohorts of one or more dosing regimens in order to determine the recommended Phase 2 dose (RP2D) for subjects with relapsed or refractory AML and relapsed or refractory higher-risk myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age, at the time of signing the ICD (Informed Consent Document).
2. Subject must understand and voluntarily sign an ICD prior to any study-related assessments/procedures being conducted.
3. Relapsed or refractory AML (Acute Myeloid Leukemia) (Parts A and B) or relapsed or refractory (R/R) higher-risk MDS (Myelodysplastic Syndrome) (HR-MDS) (Part B only) as defined by World Health Organization criteria who are not suitable for other established therapies.

   1. In Part A, R/R AML
   2. In Part B, R/R AML including

      * Relapsed after allogeneic HSCT or
      * In second or later relapse or
      * Refractory to initial induction or re-induction treatment or
      * Refractory or relapse after HMA treatment (HMA failure defined as primary progression or lack of clinical benefit after a minimum of 6 cycles or unable to tolerate HMA due to toxicity) or
      * Refractory within 1 year of initial treatment (excluding those with favorable risk based on cytogenetics)
   3. In Part B, R/R HR-MDS (Revised International Prognostic Scoring System score (IPSS-R) > 3.5 points, IPSS-R calculated during screening period):

      * IPSS-R intermediate risk (in combination with more than 10% bone marrow blasts or poor or very poor IPSS-R cytogenetic risk) or
      * IPSS-R high or
      * IPSS-R very high risk
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2.
5. At least 4 weeks (from first dose) has elapsed from donor lymphocyte infusion (DLI) without conditioning.
6. Subjects must have the following screening laboratory values:

   * Corrected serum Ca or free (ionized) serum Ca within normal limits (WNL).

     o Corrected Ca (mg/dL) = Total Ca (mg/dL) - 0.8 (albumin [g/dL] - 4)
   * Total White Blood Cell count (WBC) < 25 x 10^9/L prior to first infusion. Prior or concurrent treatment with hydroxyurea to achieve this level is allowed.
   * Potassium and magnesium within normal limits or correctable with supplements.
   * Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) or alanine aminotransferase/serum glutamate pyruvic transaminase (ALT/SGPT) ≤ 2.5 x Upper Limit of Normal (ULN).
   * Uric acid ≤ 7.5 mg/dL (446 μmol/L). Prior and/or concurrent treatment with hypouricemic agents (eg, allopurinol, rasburicase) are allowed.
   * Selected electrolytes within normal limits or correctable with supplements.
   * Serum bilirubin ≤ 1.5 x ULN (upper limit of normal).
   * Estimated serum creatinine clearance of ≥ 60 mL/min using the Cockcroft-Gault equation. Measured creatinine clearance from a 24-hour urine collection is acceptable if clinically indicated.
   * International normalized ratio (INR) < 1.5 x ULN and Partial thromboplastin time (PTT) < 1.5 x ULN.

Exclusion Criteria:

1. Subjects with acute promyelocytic leukemia (APL)
2. Subjects with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid is only required if there is clinical suspicion of CNS involvement by leukemia during screening.
3. Patients with prior autologous hematopoietic stem cell transplant who, in the investigator's judgment, have not fully recovered from the effects of the last transplant (e.g., transplant related side effects).
4. Prior allogeneic hematopoietic stem cell transplant (HSCT) with either standard or reduced intensity conditioning ≤ 6 months prior to starting CC-90009.
5. Subjects on systemic immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD).
6. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks prior to starting CC-90009, whichever is shorter. Hydroxyurea is allowed to control peripheral leukemia blasts.
7. Leukapheresis ≤ 2 weeks prior to starting CC-90009.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (6):
  - Stanford Cancer Center, Stanford, California
  - Local Institution - 105, New Haven, Connecticut
  - Local Institution - 102, Chicago, Illinois
  - Local Institution - 103, Boston, Massachusetts
  - Local Institution - 101, St Louis, Missouri
  - Local Institution - 104, Hackensack, New Jersey
- Local Institution - 201, Toronto, Ontario, Canada
- France (4):
  - Local Institution - 505, Lillie Cedex
  - Institut Paoli Calmettes, Marseille
  - Hopital Lyon Sud, Pierre-Bénite
  - Local Institution - 502, Toulouse
- Norway (2):
  - Local Institution - 700, Bergen
  - Local Institution - 701, Oslo
- Spain (6):
  - Local Institution - 603, Badalona
  - Local Institution - 602, Barcelona
  - Local Institution - 604, Madrid
  - Local Institution - 605, Pamplona
  - Local Institution - 601, Salamanca
  - Local Institution - 600, Valencia
- Local Institution - 301, Oxford, United Kingdom

REFERENCES:
- [Derived] Surka C, Jin L, Mbong N, Lu CC, Jang IS, Rychak E, Mendy D, Clayton T, Tindall E, Hsu C, Fontanillo C, Tran E, Contreras A, Ng SWK, Matyskiela M, Wang K, Chamberlain P, Cathers B, Carmichael J, Hansen J, Wang JCY, Minden MD, Fan J, Pierce DW, Pourdehnad M, Rolfe M, Lopez-Girona A, Dick JE, Lu G. CC-90009, a novel cereblon E3 ligase modulator, targets acute myeloid leukemia blasts and leukemia stem cells. Blood. 2021 Feb 4;137(5):661-677. doi: 10.1182/blood.2020008676. PMID 33197925
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - 0.3 mg: Part A - CC-90009 QD 0.3 mg (Days 1 - 5 of 28)
- Part A - 0.6 mg: Part A - CC-90009 QD 0.6 mg (Days 1 - 5 of 28)
- Part A - 1.2 mg: Part A - CC-90009 QD 1.2 mg (Days 1 - 5 of 28)
- Part A - 2.4 mg: Part A - 2.4 mg (Days 1 - 5 of 28)
- Part A - 3.0 mg: Part A - CC-90009 QD 3.0 mg (Days 1 - 5 of 28)
- Part A - 3.6 mg: Part A - CC-90009 QD 3.6 mg (Days 1 - 5 of 28)
- Part A - 3.6 mg + DEX: Part A - CC-90009 QD 3.6 mg + Dexamethasone 10 mg IV (Days 1 - 5 of 28)
- Part A - 4.5 mg: Part A - CC-90009 daily (QD) 4.5 mg (Days 1 - 5 of 28)
- Part A - 3.6 mg (Days 1 - 7 of 28): Part A - CC-90009 QD 3.6 mg (Days 1 - 7 of 28)
- Part A - 3.0 mg (Days 1- 10 of 28): Part A - CC-90009 QD 3.0 mg (Days 1- 10 of 28)
- Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28): Part A - CC-90009 daily (QD) 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28)
- Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28): Part A - CC-90009 daily (QD) 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28)
- Part B - AML 3.6 mg + DEX: Part B - 3.6 mg + DEX (Days 1 - 5 of 28)
- Part B - MDS 3.6 mg + DEX: Part B - MDS CC-90009 3.6 mg + Dexamethasone (Days 1 - 5 of 28)
- Part B - AML 2.4 mg: Part B - AML CC-90009 2.4 mg (Days 1 - 7 of 28)
- Part B - AML 3.0 mg: Part B - 3.0 mg (Days 1 - 7 of 28)
- Part B - MDS 3.0 mg: Part B - MDS 3.0 mg (Days 1 - 7 of 28)
Period: Overall Study
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Started | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 8 | 9 | 1
Not completed — other reasons | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 0
Not completed — Progressive Disease | 2 | 1 | 0 | 4 | 3 | 0 | 4 | 1 | 0 | 2 | 3 | 2 | 1 | 0 | 2 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 3 | 4 | 1 | 0 | 1 | 3 | 0 | 2 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (8.49) | 70.0 (11.31) | 60.0 (8.49) | 69.6 (8.81) | 62.2 (10.47) | 71.3 (6.81) | 59.0 (20.20) | 57.3 (17.76) | 66.0 (7.05) | 53.1 (18.20) | 64.3 (15.28) | 63.0 (17.01) | 63.3 (4.43) | 76.5 (2.12) | 66.0 (11.05) | 75.1 (7.25) | 53.0 (NA) — Unable to calculate standard deviation with 1 participant only | 63.9 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 2 | 1 | 1 | 3 | 3 | 4 | 1 | 3 | 4 | 0 | 2 | 4 | 0 | 33
  Male | 1 | 0 | 2 | 5 | 13 | 2 | 7 | 4 | 4 | 5 | 2 | 4 | 4 | 2 | 7 | 5 | 1 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 9
  Not Hispanic or Latino | 1 | 2 | 2 | 7 | 14 | 3 | 7 | 6 | 7 | 9 | 3 | 6 | 7 | 2 | 6 | 7 | 1 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  White | 2 | 1 | 1 | 3 | 13 | 3 | 6 | 6 | 7 | 8 | 2 | 5 | 6 | 2 | 6 | 7 | 1 | 79
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLTs)
Description: A participant evaluable for DLT is defined as one that: Has received at least 80% of the total planned Cycle 1 dose (eg, ≥ 4 CC-90009 doses for the Days 1-5 schedule to be completed on or before Day 10, ≥ 6 CC-90009 doses for the Days 1- 7 schedule to be completed on or before Day 10, ≥8 doses by Day 14 for the Days 1-10 schedule, or ≥ 5 doses by Day 14 for the D1-3/D8-10 schedule) of CC-90009 during Cycle 1 without experiencing a DLT, Or; Experienced a DLT after receiving at least one dose (or fraction thereof) of CC-90009 in part A.
Time Frame: From first dose to at least 28 days and up to 42 days post first dose (Up to 42 days)
Population: All treated participants in dose escalation (Part A)
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28)
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7
Participants | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 1

2. Secondary Outcome: Non-Tolerated Dose (NTD) of CC-90009
Description: The NTD is defined as a dose level at which 2 or more of up to 6 evaluable participants in any dose cohort experience a DLT in Cycle 1 during dose escalation (Part A)
Time Frame: From first dose to at least 28 days and up to 42 days post first dose (Up to 42 days)
Population: All treated participants in dose escalation (Part A)
Measure: Number; unit: mg
Groups:
- Dose Escalation (Part A): Dose Escalation (Part A) of CC-90009
Arm/Group | Dose Escalation (Part A)
Number analyzed (Participants) | 72
mg | 4.5

3. Secondary Outcome: Maximum Tolerated Dose (MTD) of CC-90009
Description: The MTD is defined as the last dose level(s) below the NTD with 0 or 1 out of 6 evaluable participants experiencing a DLT in Cycle 1 during dose escalation (part A).
Time Frame: From first dose to at least 28 days and up to 42 days post first dose (Up to 42 days)
Population: All treated participants in dose escalation (Part A)
Measure: Number; unit: mg
Arm/Group | Dose Escalation (Part A)
Number analyzed (Participants) | 72
mg | 3.6

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Treatment-emergent adverse events (TEAEs) are defined as any AEs that begin on or after the start of study drug through 28 days after the last dose of study drug or serious AEs that are suspected of being related to study drug.
Time Frame: From first dose until 28 days post last dose (Up to 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Part B - MDS 3.6 mg + DEX: Part B - MDS 3.6 mg + DEX (Days 1 - 5 of 28)
- Part B - AML 2.4 mg: Part B - 2.4 mg (Days 1 - 7 of 28)
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Participants
  TEAE | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
  TEAE related to CC-90009 | 2 | 0 | 2 | 6 | 13 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 7 | 7 | 1
  Serious TEAE | 0 | 0 | 1 | 6 | 15 | 3 | 7 | 7 | 7 | 6 | 3 | 6 | 8 | 1 | 9 | 8 | 0
  Serious TEAE related to CC-90009 | 0 | 0 | 0 | 1 | 6 | 2 | 4 | 6 | 3 | 4 | 1 | 1 | 3 | 1 | 3 | 4 | 0

5. Secondary Outcome: Change From Baseline by Laboratory Test - Chemistry Parameters 1
Description: Change from baseline for chemistry laboratory parameters. Baseline = last value before start of treatment
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
g/L
  Albumin Minimum Post Baseline Value | -6.0000 (0.00000) | 0.0000 (1.41421) | -9.5000 (2.12132) | -3.9286 (3.27145) | -9.8000 (6.82642) | -11.3333 (2.51661) | -7.7500 (4.65219) | -12.2857 (6.29058) | -9.8571 (4.74091) | -9.3333 (3.57071) | -7.6667 (4.04145) | -6.5714 (3.99404) | -9.6250 (5.73056) | -14.5000 (12.02082) | -4.2778 (4.29062) | -5.9444 (2.55495) | -2.0000 (NA) — SD not calculated due to insufficient number of participants
  Albumin Maximum Post Baseline Value | 6.5000 (4.94975) | 10.5000 (7.77817) | 2.0000 (2.82843) | 4.2143 (3.16039) | 1.7333 (7.43031) | 7.6667 (5.13160) | 4.6250 (3.20435) | 3.4286 (3.69040) | 2.7143 (4.23140) | 2.8889 (3.75648) | 4.3333 (1.52753) | 3.4286 (2.93582) | 1.6250 (3.11391) | 0.5000 (4.94975) | 5.0444 (2.56861) | 4.0778 (3.25645) | 8.0000 (NA) — SD not calculated due to insufficient number of participants
  Protein Minimum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 8 | 8 | 1
  Protein Minimum Post Baseline Value | -11.0000 (5.65685) | -1.0000 (4.24264) | -13.0000 (1.41421) | -9.7143 (5.31395) | -12.8667 (4.43793) | -20.6667 (9.50438) | -12.2500 (5.39179) | -16.5714 (3.86683) | -18.4286 (5.19157) | -16.8889 (8.00694) | -12.0000 (3.60555) | -9.8571 (4.84522) | -16.7500 (8.11964) | -16.0000 (8.48528) | -10.6750 (3.67064) | -10.7500 (5.06388) | -3.0000 (NA) — SD not calculated due to insufficient number of participants
  Protein Maximum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 8 | 8 | 1
  Protein Maximum Post Baseline Value | 8.5000 (6.36396) | 13.5000 (7.77817) | 4.5000 (4.94975) | 5.7143 (6.10230) | 122.8667 (449.87615) | 7.0000 (6.08276) | 6.8750 (7.07990) | 4.2857 (5.25085) | 2.1429 (4.41318) | 4.2222 (6.86982) | 7.3333 (4.93288) | 6.0000 (2.94392) | 0.1250 (4.61171) | 4.5000 (2.12132) | 5.7375 (4.72469) | 5.6250 (5.01248) | 13.0000 (NA) — SD not calculated due to insufficient number of participants

6. Secondary Outcome: Change From Baseline by Laboratory Test - Chemistry Parameters 2
Description: Change from baseline for chemistry laboratory parameters. Baseline = last value before start of treatment
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
U/L
  Alkaline Phosphatase (Serum) Minimum Post Baseline Value | -23.0000 (16.97056) | -4.5000 (4.94975) | -26.7500 (20.85965) | 4.1429 (57.68428) | -27.9333 (25.48520) | -29.6667 (40.27820) | -55.6250 (101.06142) | -52.4286 (66.26678) | -57.8571 (68.82448) | -15.6667 (19.00000) | -4.0000 (3.60555) | -17.7143 (18.56264) | -18.6250 (10.50085) | -14.5000 (0.70711) | -25.5222 (51.20380) | -9.7778 (12.80408) | -12.0000 (NA) — SD not calculated due to insufficient number of participants
  Alkaline Phosphatase (Serum) Maximum Post Baseline Value | 4.5000 (9.19239) | 85.5000 (67.17514) | 14.2500 (13.08148) | 104.7143 (135.05766) | 49.4000 (45.70839) | 78.0000 (84.43341) | 95.7500 (123.57733) | 72.7143 (80.35487) | 138.8571 (239.39815) | 27.2222 (24.80815) | 294.3333 (402.47898) | 47.8571 (39.29982) | 19.2500 (18.85092) | 34.0000 (8.48528) | 49.3333 (59.21571) | 39.5556 (45.42057) | 24.0000 (NA) — SD not calculated due to insufficient number of participants
  Alanine Aminotransferase (Serum) Minimum Post Baseline Value | -6.0000 (5.65685) | -5.0000 (7.07107) | -12.7500 (8.13173) | -1.6429 (20.22110) | -11.6000 (16.83024) | 11.26943 (14.0000) | -3.3750 (11.17315) | -3.5714 (21.62450) | -1.5714 (2.29907) | -0.3333 (9.44722) | -22.0000 (20.07486) | -6.1429 (5.66947) | -12.6250 (15.17458) | -8.5000 (2.12132) | -2.8889 (5.81903) | -10.6667 (13.03840) | 1.0000 (NA) — SD not calculated due to insufficient number of participants
  Alanine Aminotransferase (Serum) Maximum Post Baseline Value | 11.5000 (6.36396) | 23.5000 (13.43503) | 24.2500 (7.42462) | 63.7857 (42.38500) | 73.8000 (71.88304) | 38.0000 (14.10674) | 117.7500 (64.07083) | 150.1429 (136.43488) | 95.1429 (46.31209) | 145.8889 (141.73077) | 293.0000 (309.51090) | 49.7143 (40.91338) | 70.0000 (110.09476) | 38.0000 (11.31371) | 78.4444 (89.89176) | 52.8889 (40.26613) | 349.0000 (NA) — SD not calculated due to insufficient number of participants
  Amylase (Serum) Minimum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 6 | 11 | 1 | 6 | 4 | 4 | 4 | 3 | 6 | 3 | 2 | 6 | 5 | 1
  Amylase (Serum) Minimum Post Baseline Value | -8.0000 (8.48528) | 60.0000 (89.09545) | -7.0000 (8.48528) | 0.8333 (15.81666) | 7.6364 (28.68893) | -4.0000 (NA) — SD not calculated due to insufficient number of participants | 12.0000 (20.34699) | -12.7500 (19.60230) | 0.0000 (23.93045) | 0.7500 (14.31491) | -13.3333 (28.36077) | 20.1667 (26.11832) | -4.0000 (3.00000) | -4.0000 (8.48528) | 19.6667 (46.16348) | -18.8000 (25.50882) | 13.0000 (NA) — SD not calculated due to insufficient number of participants
  Amylase (Serum) Maximum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 6 | 11 | 1 | 6 | 4 | 4 | 4 | 3 | 6 | 3 | 2 | 6 | 5 | 1
  Amylase (Serum) Maximum Post Baseline Value | 2.5000 (3.53553) | 207.0000 (282.84271) | 1.5000 (3.53553) | 1.8333 (15.71517) | 14.4545 (27.40206) | 21.0000 (NA) — SD not calculated due to insufficient number of participants | 12.1667 (20.28218) | 17.0000 (18.67262) | 8.5000 (21.56386) | 4.5000 (10.84743) | 2.6667 (45.08141) | 22.0000 (24.23221) | -4.0000 (3.00000) | 8.0000 (7.07107) | 20.0000 (46.32926) | -11.6000 (27.71823) | 17.0000 (NA) — SD not calculated due to insufficient number of participants
  Aspartate Aminotransferase (Serum) Minimum Post Baseline Value | -4.5000 (0.70711) | -1.5000 (2.12132) | -9.7500 (2.47487) | -1.8571 (4.63424) | -7.8667 (10.94706) | -23.3333 (14.57166) | -9.8750 (13.37842) | -10.2857 (12.41926) | -4.2857 (6.23737) | -1.6667 (6.80074) | -7.6667 (7.09460) | -8.1429 (9.09997) | -8.9 (7.26) | -7.5 (0.71) | -3.6667 (5.02494) | -4.6667 (5.70088) | -8.0000 (NA) — SD not calculated due to insufficient number of participants
  Aspartate Aminotransferase (Serum) Maximum Post Baseline Value | 7.5000 (2.12132) | 17.5000 (3.53553) | 16.2500 (6.01041) | 84.1429 (82.69105) | 143.3333 (353.35629) | 55.3333 (10.96966) | 95.7500 (105.06019) | 151.2857 (282.47992) | 72.5714 (57.86149) | 74.1111 (71.85479) | 280.3333 (324.62491) | 32.8571 (36.56241) | 81.5 (171.64) | 25.0 (2.83) | 63.2222 (92.19650) | 30.0000 (23.53189) | 299.0000 (NA) — SD not calculated due to insufficient number of participants

7. Secondary Outcome: Change From Baseline by Laboratory Test - Chemistry Parameters 3
Description: Change from baseline for chemistry laboratory parameters. Baseline = last value before start of treatment
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
mmol/L
  Bicarbonate (Serum) Minimum Post Baseline Value: number analyzed (Participants) | 1 | 0 | 0 | 4 | 7 | 1 | 4 | 3 | 4 | 8 | 3 | 4 | 6 | 0 | 4 | 5 | 0
  Bicarbonate (Serum) Minimum Post Baseline Value | 0.0000 (NA) — SD not calculated due to insufficient number of participants |  |  | -8.5000 (1.29099) | -7.5143 (3.49401) | -3.0000 (NA) — SD not calculated due to insufficient number of participants | -4.0250 (2.30416) | -5.0333 (1.00167) | -11.8675 (9.78371) | -7.4500 (3.97492) | -4.1000 (1.90526) | -5.8750 (2.32289) | -3.87 (3.308) |  | -3.3500 (2.59936) | -4.6800 (1.73551) |
  Bicarbonate (Serum) Maximum Post Baseline Value: number analyzed (Participants) | 1 | 0 | 0 | 4 | 7 | 1 | 4 | 3 | 4 | 8 | 3 | 4 | 6 | 0 | 4 | 5 | 0
  Bicarbonate (Serum) Maximum Post Baseline Value | 5.0000 (NA) — SD not calculated due to insufficient number of participants |  |  | 1.0000 (1.41421) | 2.1857 (2.18893) | -2.0000 (NA) — SD not calculated due to insufficient number of participants | 6.8250 (4.57265) | 2.3000 (1.75784) | 0.8500 (2.54755) | 3.1375 (3.55163) | 2.5667 (3.48473) | 24.8000 (47.60000) | 4.98 (3.305) |  | 3.2500 (2.62996) | 4.8800 (3.04171) |
  Calcium Corrected (Serum) Minimum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 6 | 9 | 3 | 7 | 8 | 2 | 5 | 5 | 0
  Calcium Corrected (Serum) Minimum Post Baseline Value | -0.1250 (0.02121) | -0.1350 (0.01414) | -0.2350 (0.14849) | -0.4614 (0.18940) | -0.4643 (0.19304) | -0.4750 (0.30311) | -0.6106 (0.29461) | -0.5136 (0.13300) | -0.6050 (0.22163) | -0.4367 (0.10256) | -0.5350 (0.11034) | -0.4500 (0.22224) | -0.4425 (0.14071) | -0.6450 (0.13435) | -0.4800 (0.12119) | -0.4240 (0.14415) |
  Calcium Corrected (Serum) Maximum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 6 | 9 | 3 | 7 | 8 | 2 | 5 | 5 | 0
  Calcium Corrected (Serum) Maximum Post Baseline Value | 0.1550 (0.00707) | 0.1475 (0.10253) | 0.2025 (0.21567) | 0.1064 (0.20428) | 0.1757 (0.11539) | 0.0917 (0.14216) | 0.1431 (0.16641) | 0.1157 (0.13148) | 0.2175 (0.07777) | 0.1417 (0.20335) | -0.0283 (0.11361) | 0.0957 (0.11002) | 0.1063 (0.10374) | 0.0300 (0.19799) | 0.0740 (0.09397) | 0.1630 (0.06676) |
  Calcium, Ionized (Blood) (mmol/L) Minimum Post Baseline Value: number analyzed (Participants) | 1 | 0 | 1 | 3 | 9 | 1 | 5 | 6 | 7 | 9 | 0 | 7 | 7 | 2 | 5 | 5 | 1
  Calcium, Ionized (Blood) (mmol/L) Minimum Post Baseline Value | 0.0225 (NA) — SD not calculated due to insufficient number of participants |  | -0.2225 (NA) — SD not calculated due to insufficient number of participants | -0.2033 (0.05774) | -0.1558 (0.27691) | -0.3700 (NA) — SD not calculated due to insufficient number of participants | -0.2220 (0.08831) | -0.3242 (0.33363) | -0.3950 (0.23569) | -0.2364 (0.10346) |  | -0.2696 (0.12539) | -0.1971 (0.05376) | -0.5275 (0.20506) | -0.1815 (0.10910) | -0.0820 (0.67998) | -0.0925 (NA) — SD not calculated due to insufficient number of participants
  Calcium, Ionized (Blood) (mmol/L) Maximum Post Baseline Value: number analyzed (Participants) | 1 | 0 | 1 | 3 | 9 | 1 | 5 | 6 | 7 | 9 | 0 | 7 | 7 | 2 | 5 | 5 | 1
  Calcium, Ionized (Blood) (mmol/L) Maximum Post Baseline Value | 0.0225 (NA) — SD not calculated due to insufficient number of participants |  | 0.0150 (NA) — SD not calculated due to insufficient number of participants | -0.0350 (0.09124) | 0.3386 (0.42193) | -0.0200 (NA) — SD not calculated due to insufficient number of participants | 0.2740 (0.44510) | -0.0138 (0.10585) | 17.3332 (45.22988) | 0.0592 (0.09937) |  | 0.0989 (0.11111) | 0.0643 (0.08204) | -0.0438 (0.10076) | 0.0575 (0.13083) | 0.5025 (0.62937) | 0.0725 (NA) — SD not calculated due to insufficient number of participants
  Chloride (Serum) Minimum Post Baseline Value | -4.5000 (0.70711) | -9.5000 (4.94975) | -5.0000 (1.41421) | -4.4286 (2.37045) | -10.1333 (24.80169) | -5.0000 (5.29150) | -7.3750 (4.77905) | -5.5714 (2.93582) | -15.4286 (29.94916) | -5.1111 (3.48010) | -3.0000 (1.00000) | -5.4286 (2.82000) | -3.1250 (4.58063) | -4.5000 (0.70711) | -4.1889 (3.81394) | -14.4444 (21.11345) | -8.0000 (NA) — SD not calculated due to insufficient number of participants
  Chloride (Serum) Maximum Post Baseline Value | 3.5000 (0.70711) | 0.5000 (3.53553) | 6.5000 (3.53553) | 5.0000 (3.36650) | 9.4000 (8.64209) | 11.6667 (3.05505) | 5.0000 (2.56348) | 5.4286 (3.40867) | 10.7143 (7.99405) | 5.1111 (3.10018) | 4.3333 (1.15470) | 5.4286 (4.57738) | 6.0000 (5.58058) | 6.0000 (2.82843) | 3.6333 (3.39264) | 6.0000 (8.06226) | 0.0000 (NA) — SD not calculated due to insufficient number of participants
  Carbon Dioxide (Plasma) Minimum Post Baseline Value: number analyzed (Participants) | 1 | 2 | 2 | 3 | 11 | 3 | 6 | 5 | 4 | 7 | 2 | 3 | 5 | 2 | 6 | 4 | 1
  Carbon Dioxide (Plasma) Minimum Post Baseline Value | -6.00 (NA) — SD not calculated due to insufficient number of participants | -3.00 (0.000) | -4.00 (4.243) | -7.83 (5.393) | -6.15 (2.716) | -7.33 (2.082) | -8.92 (5.788) | -13.12 (7.367) | -10.18 (4.032) | -9.59 (4.171) | -3.00 (2.404) | -7.67 (1.528) | -5.5600 (6.65004) | -8.0000 (4.24264) | -5.2333 (4.26224) | -5.5000 (2.38048) | -9.0000 (NA) — SD not calculated due to insufficient number of participants
  Carbon Dioxide (Plasma) Maximum Post Baseline Value: number analyzed (Participants) | 1 | 2 | 2 | 3 | 11 | 3 | 6 | 5 | 4 | 7 | 2 | 3 | 5 | 2 | 6 | 4 | 1
  Carbon Dioxide (Plasma) Maximum Post Baseline Value | 5.00 (NA) — SD not calculated due to insufficient number of participants | 4.00 (0.000) | 7.00 (2.828) | 5.50 (7.089) | 7.02 (8.784) | 2.67 (2.082) | 4.88 (5.841) | 2.06 (3.531) | 1.25 (3.304) | 3.93 (3.622) | 25.20 (5.374) | 0.67 (2.082) | 3.5200 (4.35282) | 2.5000 (3.53553) | 1.7500 (1.99374) | 3.0000 (2.58199) | 1.0000 (NA) — SD not calculated due to insufficient number of participants
  Glucose (Serum Fasting) Minimum Post Baseline Value | -0.7333 (0.80151) | -1.7205 (0.78489) | -2.1229 (0.80451) | -1.7822 (1.22271) | -1.9303 (1.73875) | -2.0165 (1.28292) | -1.7267 (1.12065) | -1.2917 (2.58471) | -0.7142 (1.10594) | -0.3899 (1.35398) | -0.9662 (0.69337) | -1.2026 (1.14734) | -2.7784 (3.30908) | -1.6650 (2.04071) | -2.0524 (1.98069) | -3.8089 (4.81888) | -0.7770 (NA) — SD not calculated due to insufficient number of participants
  Glucose (Serum Fasting) Maximum Post Baseline Value | 2.6098 (0.15521) | 2.4698 (2.62938) | 5.8136 (2.02109) | 2.4246 (2.08954) | 3.0881 (2.37534) | 5.9755 (5.04847) | 6.6410 (12.50771) | 6.6956 (4.61321) | 4.2604 (3.84923) | 4.0611 (2.96891) | 3.3685 (1.95592) | 5.6909 (4.20310) | 4.5039 (5.49686) | 5.49686 (2.27618) | 2.5520 (3.08923) | 3.0482 (7.55874) | 3.4410 (NA) — SD not calculated due to insufficient number of participants
  Potassium (Serum) Minimum Post Baseline Value | -0.5500 (0.07071) | -0.6500 (0.63640) | -0.6750 (0.53033) | -0.9457 (0.75540) | -0.7000 (0.56821) | -0.6667 (0.40415) | -0.8750 (0.58737) | -0.8214 (0.34139) | -1.0571 (0.29921) | -0.8667 (0.53852) | -1.1000 (0.36056) | -0.7857 (0.29681) | -0.6875 (0.58661) | -0.7500 (0.35355) | -0.5000 (0.30000) | -0.7778 (0.40242) | -0.7000 (NA) — SD not calculated due to insufficient number of participants
  Potassium (Serum) Maximum Post Baseline Value | 0.5000 (0.28284) | 0.5000 (0.28284) | 0.2250 (0.17678) | 0.7286 (0.47859) | 0.5400 (0.35416) | 0.7000 (0.98489) | 0.4625 (0.27223) | 0.6071 (0.32968) | 0.5857 (0.55806) | 0.3111 (0.32189) | 0.4000 (0.43589) | 0.7286 (0.85579) | 0.7125 (0.44219) | 0.5500 (0.49497) | 0.4933 (0.52192) | 15.2000 (44.25113) | 0.2000 (NA) — SD not calculated due to insufficient number of participants
  Magnesium (Serum) Minimum Post Baseline Value | -0.1678 (0.05339) | -0.0822 (0.11625) | -0.1747 (0.04359) | -0.1325 (0.09877) | -0.1434 (0.15976) | -0.0685 (0.06278) | -0.1816 (0.11047) | -0.1621 (0.12041) | -0.1554 (0.13947) | -0.1364 (0.11191) | -0.1742 (0.11591) | -0.1289 (0.12833) | -0.0969 (0.07597) | -0.0822 (0.05812) | -0.0995 (0.07483) | -0.0616 (0.06859) | -0.1233 (NA) — SD not calculated due to insufficient number of participants
  Magnesium (Serum) Maximum Post Baseline Value | 0.0661 (0.02277) | 0.2466 (0.29062) | 0.0514 (0.07266) | 0.3527 (0.17041) | 0.2818 (0.14292) | 0.2466 (0.12330) | 0.1397 (0.15729) | 0.2115 (0.17599) | 0.2198 (0.21791) | 0.2259 (0.11524) | 0.1604 (0.12659) | 0.5257 (0.79291) | 0.2620 (0.24586) | 0.7213 (0.26447) | 0.2454 (0.16916) | 0.2256 (0.12779) | 0.1644 (NA) — SD not calculated due to insufficient number of participants
  Phosphate (Serum) Minimum Post Baseline Value | -0.4757 (0.14948) | -0.0485 (0.06852) | -0.3069 (0.06852) | -0.6302 (0.26517) | -0.5801 (0.28215) | -0.7752 (0.43455) | -0.6085 (0.28717) | -0.5723 (0.25444) | -0.4597 (0.38489) | -0.6305 (0.25010) | -1.0614 (0.37317) | -0.7058 (0.31457) | -0.4598 (0.50333) | -0.5168 (0.31975) | -0.4614 (0.29484) | -0.2159 (0.25466) | -0.3553 (NA) — SD not calculated due to insufficient number of participants
  Phosphate (Serum) Maximum Post Baseline Value | 0.1396 (0.01471) | 0.3715 (0.11420) | 0.4684 (0.38827) | 0.7003 (0.49600) | 0.7392 (0.61769) | 0.5276 (0.57448) | 0.6354 (0.51976) | 1.1399 (0.73804) | 0.8597 (0.91607) | 0.3119 (0.55165) | 0.0392 (0.12539) | 0.6580 (0.48893) | 0.8600 (0.82275) | 0.4684 (0.29691) | 0.6059 (0.33589) | 0.4636 (0.35631) | 0.0646 (NA) — SD not calculated due to insufficient number of participants
  Sodium (Serum) Minimum Post Baseline Value | -7.0000 (2.82843) | -4.0000 (1.41421) | -7.5000 (4.94975) | -5.4286 (2.50713) | -7.1333 (7.98093) | -4.0000 (3.60555) | -6.1250 (2.53194) | -6.4286 (2.22539) | -5.0000 (1.15470) | -6.8889 (2.84800) | -7.0000 (1.00000) | -5.5714 (2.69921) | -2.6250 (3.42000) | -8.5000 (2.12132) | -4.4111 (2.97844) | -5.2222 (3.49205) | -12.0000 (NA) — SD not calculated due to insufficient number of participants
  Sodium (Serum) Maximum Post Baseline Value | 1.0000 (0.00000) | 2.5000 (2.12132) | 3.5000 (0.70711) | 2.7143 (3.25137) | 4.6667 (4.13464) | 5.3333 (6.50641) | 3.3750 (5.65528) | 2.4286 (3.10146) | 5.7143 (6.04743) | 1.6667 (1.58114) | 1.6667 (2.08167) | 2.5714 (0.97590) | 4.5000 (4.47214) | 0.0000 (1.41421) | 2.6778 (2.53662) | 3.8889 (2.66667) | -1.0000 (NA) — SD not calculated due to insufficient number of participants
  Blood Urea Nitrogen (Serum) Minimum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 6 | 7 | 8 | 3 | 7 | 8 | 2 | 7 | 7 | 1
  Blood Urea Nitrogen (Serum) Minimum Post Baseline Value | -2.1640 (1.04086) | -0.8925 (1.76706) | -2.1420 (1.51462) | -1.9180 (1.23345) | -1.4420 (1.63613) | -1.7850 (0.94453) | -1.6767 (1.92439) | -1.3615 (1.87780) | -1.3589 (1.65079) | -1.1995 (2.01204) | -1.8114 (0.77173) | -0.8080 (1.44364) | -0.2616 (1.46975) | -3.7485 (1.26219) | -1.4423 (2.08076) | -0.9405 (1.10505) | 0.0000 (NA) — SD not calculated due to insufficient number of participants
  Blood Urea Nitrogen (Serum) Maximum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 6 | 7 | 8 | 3 | 7 | 8 | 2 | 7 | 7 | 1
  Blood Urea Nitrogen (Serum) Maximum Post Baseline Value | 2.4780 (0.53457) | 4.9980 (2.01950) | 5.1765 (0.75731) | 6.8120 (6.77422) | 8.3157 (4.35216) | 9.5200 (8.51827) | 9.7553 (5.39524) | 13.6523 (8.34637) | 14.8533 (9.94930) | 11.0090 (3.89546) | 10.5890 (13.37754) | 10.5656 (5.62941) | 10.1050 (7.49087) | 11.4240 (0.50487) | 7.6687 (2.92428) | 8.1828 (4.82377) | 8.5680 (NA) — SD not calculated due to insufficient number of participants

8. Secondary Outcome: Change From Baseline for Vital Signs by Test - Parameters 1
Description: Change from Baseline for Vital Signs Parameters. Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
mmHg
  Systolic Blood Pressure Minimum Post Baseline Value | -18.5 (3.54) | -15.0 (2.83) | -19.5 (13.44) | -37.0 (16.73) | -27.9 (14.65) | -54.0 (16.64) | -27.8 (13.58) | -35.1 (16.20) | -29.1 (10.46) | -23.0 (12.27) | -36.7 (23.07) | -17.1 (10.90) | -22.8 (12.79) | -10.0 (11.31) | -27.3 (16.65) | -29.1 (18.20) | -31.0 (NA) — SD not calculated due to insufficient number of participants
  Systolic Blood Pressure Maximum Post Baseline Value | 23.0 (0.00) | 33.0 (0.00) | 18.5 (7.78) | 18.6 (20.86) | 22.1 (13.36) | 9.3 (7.77) | 29.5 (16.25) | 26.1 (10.57) | 25.4 (11.25) | 30.8 (18.08) | 20.0 (8.54) | 29.0 (8.33) | 25.3 (12.68) | 45.5 (23.33) | 24.4 (9.50) | 27.3 (21.51) | 26.0 (NA) — SD not calculated due to insufficient number of participants
  Diastolic Blood Pressure Minimum Post Baseline Value | -7.0 (7.07) | -2.0 (7.07) | -18.0 (19.80) | -16.7 (6.65) | -16.8 (7.18) | -22.7 (9.87) | -17.8 (6.36) | -17.3 (8.44) | -19.1 (8.43) | -15.0 (12.87) | -25.7 (11.55) | -14.9 (10.79) | -16.6 (11.90) | -13.0 (14.14) | -17.2 (7.60) | -19.1 (11.47) | -10.0 (NA) — SD not calculated due to insufficient number of participants
  Diastolic Blood Pressure Maximum Post Baseline Value | 23.0 (0.00) | 33.0 (4.24) | 12.5 (6.36) | 16.6 (1.90) | 17.4 (13.29) | 10.3 (2.08) | 22.6 (9.96) | 17.7 (8.26) | 18.3 (9.43) | 23.6 (9.70) | 15.0 (3.46) | 19.4 (13.72) | 17.9 (8.37) | 20.0 (9.90) | 16.9 (11.54) | 14.3 (16.01) | 26.0 (NA) — SD not calculated due to insufficient number of participants

9. Secondary Outcome: Change From Baseline for Vital Signs by Test - Parameters 2
Description: Change from Baseline for Vital Signs Parameters. Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
beats/min
  Pulse Minimum Post Baseline Value | -15.5 (4.95) | -6.0 (5.66) | -21.5 (10.61) | -9.7 (13.41) | -14.1 (10.85) | -23.0 (12.12) | -14.0 (8.47) | -14.7 (10.34) | -25.1 (14.10) | -18.4 (10.43) | -22.7 (9.50) | -24.7 (19.90) | -15.6 (9.59) | -11.0 (8.49) | -21.9 (8.10) | -11.8 (9.58) | -20.0 (NA) — SD not calculated due to insufficient number of participants
  Pulse Maximum Post Baseline Value | 29.0 (9.90) | 28.0 (8.49) | 17.0 (18.38) | 27.7 (24.98) | 32.0 (12.10) | 14.0 (18.25) | 38.9 (16.86) | 23.9 (12.33) | 30.6 (16.53) | 26.3 (22.84) | 28.0 (19.00) | 22.1 (10.99) | 29.4 (12.69) | 43.5 (13.44) | 21.7 (21.82) | 25.3 (14.93) | 32.0 (NA) — SD not calculated due to insufficient number of participants
  Respiration Minimum Post Baseline Value | -1.0 (1.41) | -3.0 (1.41) | -2.0 (0.00) | -1.0 (1.73) | -1.9 (1.39) | -2.3 (2.52) | -2.4 (2.97) | -2.4 (2.57) | -4.9 (1.95) | -1.1 (1.36) | -1.7 (2.08) | -2.9 (2.79) | -2.8 (3.41) | -3.5 (2.12) | -2.4 (1.59) | -3.3 (2.65) | -2.0 (NA) — SD not calculated due to insufficient number of participants
  Respiration Maximum Post Baseline Value | 2.0 (2.83) | 3.0 (3.0) | 4.0 (2.83) | 2.9 (1.68) | 5.0 (5.15) | 4.0 (2.00) | 3.9 (2.64) | 4.7 (3.82) | 2.9 (1.07) | 3.4 (3.36) | 3.7 (0.58) | 5.3 (4.11) | 3.3 (3.58) | 2.0 (0.00) | 3.9 (6.95) | 1.6 (1.42) | 2.0 (NA) — SD not calculated due to insufficient number of participants

10. Secondary Outcome: Change From Baseline for Vital Signs by Test - Parameters 3
Description: Change from Baseline for Vital Signs Parameters. Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Celsius
  Temperature Minimum Post Baseline Value | -0.15 (0.354) | -0.45 (0.212) | -0.25 (0.354) | -0.50 (0.392) | -0.77 (0.443) | -1.47 (1.686) | -0.61 (0.340) | -0.76 (0.395) | -1.69 (0.830) | -1.08 (0.499) | -0.50 (0.300) | -1.16 (0.678) | -0.99 (0.511) | -0.55 (0.354) | -0.74 (0.456) | -3.31 (6.473) | -0.60 (NA) — SD not calculated due to insufficient number of participants
  Temperature Maximum Post Baseline Value | 0.65 (0.778) | 0.65 (0.212) | 0.80 (0.566) | 0.77 (0.591) | 0.93 (0.704) | -0.03 (0.513) | 0.86 (0.657) | 1.67 (1.378) | 0.73 (0.647) | 0.39 (0.326) | 1.40 (0.866) | 0.67 (0.468) | 0.73 (0.865) | 0.25 (0.071) | 0.49 (0.607) | 6.97 (19.185) | 0.90 (NA) — SD not calculated due to insufficient number of participants

11. Secondary Outcome: Change From Baseline for Vital Signs by Test - Parameters 4
Description: Change from Baseline for Vital Signs Parameters. Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 7 | 2 | 9 | 8 | 1
Kg
  Weight Minimum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 7 | 2 | 9 | 8 | 1
  Weight Minimum Post Baseline Value | -1.20 (1.697) | -2.05 (0.495) | -4.40 (6.223) | -4.27 (3.410) | -4.51 (2.254) | -3.13 (2.928) | -5.38 (5.135) | -2.60 (3.475) | -3.86 (2.375) | -3.40 (4.310) | -3.57 (1.358) | -5.84 (1.786) | -4.37 (3.617) | -8.55 (5.303) | -2.44 (2.993) | -4.84 (3.910) | 0.00 (NA) — SD not calculated due to insufficient number of participants
  Weight Maximum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 7 | 2 | 9 | 8 | 1
  Weight Maximum Post Baseline Value | 4.00 (2.404) | 0.70 (0.424) | 2.10 (0.707) | 3.40 (4.987) | 2.19 (4.788) | 2.83 (3.539) | 2.55 (3.789) | 2.13 (2.833) | 3.89 (3.074) | 0.54 (1.415) | 1.70 (1.947) | 0.94 (2.028) | 1.27 (3.364) | 0.55 (0.778) | 0.89 (2.194) | 1.74 (3.250) | 4.60 (NA) — SD not calculated due to insufficient number of participants

12. Secondary Outcome: Change From Baseline for Electrocardiogram (ECG) by Test - Parameters 1
Description: Change from Baseline for Electrocardiogram (ECG) Parameters. Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 8 | 8 | 1
beats/min
  ECG Mean Heart Rate Minimum Post Baseline Value | -7.6667 (4.24264) | -7.3333 (3.29983) | -9.5000 (1.64992) | -12.1429 (6.43445) | -11.0667 (6.22106) | -14.6667 (16.75642) | -11.4167 (10.22563) | -17.6190 (12.60280) | -19.7619 (10.39536) | -12.6667 (7.66848) | -18.6667 (5.84047) | -14.6190 (12.27981) | -13.8333 (12.14463) | -3.5000 (8.24958) | -13.1250 (11.77560) | -15.8750 (7.08662) | -9.0000 (NA) — SD not calculated due to insufficient number of participants
  ECG Mean Heart Rate Maximum Post Baseline Value | 34.3333 (19.79899) | 16.1667 (8.72098) | 12.0000 (2.35702) | 12.1429 (5.74088) | 14.4000 (8.57108) | 7.0000 (9.02466) | 22.3333 (13.38324) | 9.0952 (9.70627) | 16.3810 (9.12349) | 15.2222 (14.31491) | 10.0000 (12.81059) | 24.2381 (14.62331) | 12.9167 (8.59633) | 14.5000 (5.42115) | 7.5000 (7.95024) | 4.8750 (5.46253) | 22.0000 (NA) — SD not calculated due to insufficient number of participants

13. Secondary Outcome: Change From Baseline for Electrocardiogram (ECG) by Test - Parameters 2
Description: Change from Baseline for Electrocardiogram (ECG) Parameters. Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 8 | 8 | 1
msec
  RR Interval, Aggregate Minimum Post Baseline Value | -227.8333 (115.25841) | -154.1667 (60.10408) | -100.0000 (40.54079) | -88.3810 (43.76047) | -120.3111 (73.42359) | -90.3333 (130.08203) | -214.3333 (104.85455) | -87.4286 (76.34879) | -120.5714 (75.49263) | -124.4815 (110.59047) | -56.2222 (66.17513) | -172.6667 (101.57519) | -95.5833 (71.55434) | -204.1667 (102.53048) | -62.1667 (91.12036) | -49.6250 (54.53539) | -179.6667 (NA) — SD not calculated due to insufficient number of participants
  RR Interval, Aggregate Maximum Post Baseline Value | 79.1667 (37.47666) | 95.8333 (33.23402) | 101.5000 (11.07801) | 126.6190 (77.45092) | 130.0889 (103.01028) | 122.0000 (189.59694) | 155.9167 (134.00577) | 214.8571 (139.93727) | 245.8571 (205.30329) | 168.4074 (120.28609) | 189.7778 (60.61750) | 168.7619 (147.66074) | 151.7917 (121.02039) | 59.3333 (144.24978) | 136.5833 (98.81002) | 193.0000 (72.50638) | 110.3333 (NA) — SD not calculated due to insufficient number of participants
  PR Interval, Aggregate Minimum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 6 | 15 | 3 | 7 | 6 | 7 | 9 | 3 | 6 | 8 | 2 | 6 | 8 | 1
  PR Interval, Aggregate Minimum Post Baseline Value | -10.6667 (0.94281) | -17.6667 (2.82843) | -13.1667 (3.06413) | -18.3333 (9.18453) | -33.0222 (30.52672) | -12.2222 (6.16742) | -17.7619 (10.10815) | -22.1111 (9.44144) | -14.9524 (14.86785) | -26.2593 (13.96004) | -8.5556 (7.01057) | -19.5000 (15.86576) | -24.2917 (13.70950) | -25.0000 (22.62742) | -22.0000 (5.94045) | -21.2917 (15.15050) | -16.0000 (NA) — SD not calculated due to insufficient number of participants
  PR Interval, Aggregate Maximum Post Baseline Value: number analyzed (Participants) | 2 | 2 | 2 | 6 | 15 | 3 | 7 | 6 | 7 | 9 | 3 | 6 | 8 | 2 | 6 | 8 | 1
  PR Interval, Aggregate Maximum Post Baseline Value | 17.3333 (0.47140) | 11.3333 (1.41421) | 25.3333 (14.61354) | 21.1667 (16.32142) | 11.8444 (9.61387) | 13.1111 (3.35548) | 21.0952 (14.84203) | 20.8889 (18.09809) | 23.0476 (21.51866) | 8.7407 (8.21884) | 21.1111 (4.53791) | 18.0000 (17.54106) | 21.8333 (17.58697) | 13.5000 (4.94975) | 7.6667 (11.36466) | 17.9583 (12.78446) | 11.0000 (NA) — SD not calculated due to insufficient number of participants
  QRS Duration, Aggregate Minimum Post Baseline Value | -11.1667 (4.94975) | -3.6667 (5.65685) | -18.1667 (2.59272) | -6.9524 (5.68764) | -10.3333 (5.60187) | -11.4444 (2.14303) | -16.9167 (14.64582) | -13.1429 (6.33876) | -5.9048 (3.62968) | -12.5926 (5.66612) | -5.8889 (2.69430) | -10.5714 (10.26990) | -7.3750 (5.51603) | -6.6667 (0.00000) | -13.7500 (7.04802) | -9.8333 (8.09468) | -7.0000 (NA) — SD not calculated due to insufficient number of participants
  QRS Duration, Aggregate Maximum Post Baseline Value | 15.8333 (2.12132) | 11.8333 (3.53553) | 8.3333 (2.35702) | 11.3333 (6.12826) | 10.1333 (3.75182) | 10.8889 (15.25463) | 9.3333 (8.49089) | 7.0000 (6.85025) | 13.5238 (6.72711) | 7.2963 (4.94819) | 12.7778 (1.83586) | 17.2857 (17.24919) | 11.6250 (7.44170) | 14.8333 (7.77817) | 7.8750 (4.57369) | 12.2917 (5.39676) | 26.0000 (NA) — SD not calculated due to insufficient number of participants
  QT Interval, Aggregate Minimum Post Baseline Value | -47.3333 (2.82843) | -43.1667 (10.13520) | -36.0000 (2.35702) | -29.1667 (24.44400) | -35.9778 (24.63978) | -11.6667 (27.42464) | -44.8750 (22.71140) | -30.0952 (26.46361) | -36.4286 (21.44823) | -36.8889 (29.53341) | -15.7778 (18.67956) | -44.7619 (18.83526) | -37.4583 (21.83047) | -30.0000 (20.27039) | -18.2083 (28.82125) | -13.3333 (17.30033) | -43.0000 (NA) — SD not calculated due to insufficient number of participants
  QT Interval, Aggregate Maximum Post Baseline Value | 15.1667 (13.43503) | 25.8333 (6.83537) | 31.0000 (27.34146) | 33.2619 (20.14711) | 41.2889 (25.74844) | 31.0000 (33.88379) | 35.1250 (22.78257) | 49.4762 (44.13316) | 70.7143 (52.20559) | 35.7778 (19.04089) | 51.2222 (23.57101) | 40.2381 (24.11985) | 47.9167 (32.36388) | 34.5000 (30.87700) | 49.5417 (26.98144) | 57.0417 (20.03920) | 31.0000 (NA) — SD not calculated due to insufficient number of participants
  QTcB Interval, Aggregate Minimum Post Baseline Value | -26.6667 (18.85618) | -13.6667 (4.71405) | -26.1667 (7.77817) | -37.9048 (23.49288) | -26.0000 (14.11630) | -33.6667 (30.68840) | -35.9167 (12.32593) | -43.5714 (15.36315) | -23.2381 (21.81718) | -37.8519 (13.50834) | -24.3333 (12.44097) | -28.9048 (11.31160) | -27.7083 (25.60347) | -2.6667 (2.35702) | -24.5000 (19.07213) | -17.7083 (19.25059) | -19.3333 (NA) — SD not calculated due to insufficient number of participants
  QTcB Interval, Aggregate Maximum Post Baseline Value | 30.3333 (34.41253) | 29.3333 (13.67073) | 27.8333 (20.50610) | 34.0952 (14.69784) | 40.2667 (20.09154) | 40.0000 (14.16961) | 46.3333 (47.27025) | 26.5714 (12.68086) | 35.9048 (22.60999) | 30.8148 (20.01466) | 35.6667 (17.63834) | 28.6667 (14.31394) | 41.2917 (26.23728) | 57.8333 (13.90643) | 41.5000 (23.81343) | 33.5417 (2.98641) | 27.6667 (NA) — SD not calculated due to insufficient number of participants
  QTcF Interval, Aggregate Minimum Post Baseline Value | -23.3333 (15.55635) | -23.1667 (0.70711) | -24.8333 (2.59272) | -31.0000 (19.99074) | -25.9333 (17.71879) | -21.7778 (23.04665) | -32.2917 (10.84880) | -32.8095 (19.63260) | -24.1429 (17.22279) | -33.2963 (15.06047) | -15.0000 (8.37324) | -28.2381 (15.88234) | -29.5000 (23.42228) | -7.5000 (5.42115) | -18.8333 (21.34672) | -12.1250 (15.84542) | -19.0000 (NA) — SD not calculated due to insufficient number of participants
  QTcF Interval, Aggregate Maximum Post Baseline Value | 23.1667 (24.74874) | 21.3333 (8.48528) | 25.1667 (28.51997) | 30.8571 (15.99983) | 37.0000 (23.07613) | 35.5556 (15.84064) | 35.3333 (29.24120) | 30.1905 (24.71156) | 42.7143 (31.84594) | 27.1481 (13.66780) | 37.3333 (20.52911) | 25.3333 (14.23480) | 42.2500 (23.41872) | 43.5000 (8.72098) | 41.4167 (17.87767) | 36.7500 (6.69932) | 29.0000 (NA) — SD not calculated due to insufficient number of participants

14. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Number of participants with post-baseline grade increase or decrease from baseline. Grade 0=; Grade 1=; Grade 2=; Grade 3=; Grade 4=; Grade 5=; . Baseline = last value before start of treatment.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Participants
  Post Baseline Grade Increase | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 3 | 1 | 2 | 0 | 2 | 2 | 0 | 3 | 0 | 0
  Post Baseline Grade Decrease | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0

15. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) Percent Change From Baseline
Description: Left Ventricular Ejection Fraction (LVEF) percent change from baseline. Baseline = last value before start of treatment.
  Minimum Post Baseline Value=lowest value of the measured parameter is recorded after the baseline measurement.
  Maximum Post Baseline Value=highest value of the measured parameter is recorded after the baseline measurement.
Time Frame: From baseline until 28 days post last dose (Up to 25 months)
Population: All treated participants with baseline and post baseline measurements
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 1 | 4 | 7 | 1 | 4 | 3 | 5 | 3 | 2 | 4 | 2 | 2 | 3 | 3 | 1
Percent change
  Minimum Post Baseline Value | -8.1 (15.88) | 15.2 (0.88) | -3.5 (NA) — SD not calculated due to insufficient number of participants | -9.9 (17.61) | 1.8 (7.37) | -9.8 (NA) — SD not calculated due to insufficient number of participants | 3.2 (9.86) | -3.7 (8.00) | 1.8 (10.63) | 0.1 (17.54) | 2.3 (3.21) | 8.7 (10.19) | -8.3 (11.79) | 17.5 (26.66) | 5.2 (26.32) | -3.3 (8.62) | 1.0 (NA) — SD not calculated due to insufficient number of participants
  Maximum Post Baseline Value | -8.1 (15.88) | 15.2 (0.88) | -3.5 (NA) — SD not calculated due to insufficient number of participants | -9.1 (18.42) | 1.8 (7.37) | -1.6 (NA) — SD not calculated due to insufficient number of participants | 3.2 (9.86) | -3.7 (8.00) | 1.8 (10.63) | 0.1 (17.54) | 3.1 (2.11) | 8.7 (10.19) | -8.3 (11.79) | 17.5 (26.66) | 5.2 (26.32) | -3.3 (8.62) | 1.5 (NA) — SD not calculated due to insufficient number of participants

16. Secondary Outcome: Objective Response Rate (ORR)
Description: Objectve response is defined as the percent of participants whose best overall response is any type of Morphologic Complete Remission [CR] (CR, Morphologic Complete Remission with Incomplete Blood Count Recovery (CRi), Morphologic Complete Remission with Partial Hematologic Recovery (CRh), Cytogenetic Complete Remission (CRc) and Molecular Complete Remission (CRm)) or Morphologic Leukemia - Free State or partial remission. CR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; CRi=residual neutropenia < 1,000/μL, thrombocytopenia < 100,000/μL. CRh=neutrophils ≥ 500μL, platelets ≥500,000μL, blasts <5%; CRc=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; cytogenetics normal; CRm=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%, negative EMD; PR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts decrease in ≥ 50 resulting in 5 to 25%.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Percent of participants | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 6.7 [0.17 to 31.95] | 33.3 [0.84 to 90.57] | 25.0 [3.19 to 65.09] | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 57.1 [18.41 to 90.10] | 33.3 [7.49 to 70.07] | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 25.0 [3.19 to 65.09] | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR | 11.1 [0.28 to 48.25] | 0 [NA to NA] — Lower limit and upper limit not calculated due to 0 participants with ORR

17. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose to the date of death from any cause.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Months | 4.93 [2.86 to 7.00] | 8.27 [5.29 to 11.24] | 8.02 [7.10 to 8.94] | 2.79 [0.30 to 3.25] | 1.91 [1.18 to 3.45] | 8.28 [0.66 to NA] — Insufficient number of participants with events to calculate upper limit | 3.25 [0.39 to 9.76] | 1.68 [0.30 to 7.10] | 3.39 [0.89 to 3.72] | 4.70 [0.43 to 12.20] | 3.72 [1.94 to NA] — Insufficient number of participants with events to calculate upper limit | 4.18 [0.46 to 5.98] | 1.28 [0.30 to 3.75] | 7.81 [7.59 to 8.02] | 2.43 [0.39 to 5.42] | 2.30 [0.30 to 4.47] | NA [NA to NA] — Insufficient number of participants with events

18. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS is defined only for participants who achieved CR or CRi (for AML) / CR or PR (for MDS) and is measured as the interval from the date of first CR or CRi (for AML) / CR or PR (for MDS) to the date of relapse or death from any cause, whichever occurs first. CR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; CRi=residual neutropenia < 1,000 μL, thrombocytopenia < 100,000/μL. PR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts decrease in ≥ 50 resulting in 5 to 25%.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Months | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | 10.83 [8.61 to 13.05] | NA [NA to NA] — No participants with event | 2.40 [NA to NA] — Insufficient number of participants with events | NA [6.12 to NA] — Insufficient number of participants with events | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | 3.02 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event

19. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose to the date of first relapse after CR/CRi (for AML)/relapse after CR/PR(for MDS), or PD, or death resulting from any cause, whichever occurs first. CR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; CRi=residual neutropenia < 1,000 μL, thrombocytopenia < 100,000/μL. PR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts decrease in ≥ 50 resulting in 5 to 25%. PD=At least 50% decrement from maximum remission/response levels in granulocytes or platelets; Reduction in Hgb concentration by ≥ 2 g/dL; Transfusion dependence. Based on Kaplan-Meier Estimates.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Months | 1.56 [0.82 to 2.30] | 2.10 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 1.74 [0.30 to 3.25] | 1.35 [0.79 to 2.79] | 1.02 [0.66 to NA] — Insufficient number of participants with events | 1.45 [0.39 to 3.78] | 1.50 [0.30 to 7.10] | 2.60 [0.89 to 3.65] | 1.07 [0.43 to NA] — Insufficient number of participants with events | 1.94 [0.95 to 2.33] | 2.33 [0.46 to 2.93] | 1.07 [0.30 to 3.75] | 7.81 [7.59 to 8.02] | 0.90 [0.30 to 1.71] | 2.30 [0.30 to 3.75] | 1.84 [NA to NA] — Insufficient number of participants with events

20. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the interval from the date of the first dose to an event including disease progression (PD), treatment failure, relapse, or death from any cause, whichever occurs first. PD=At least 50% decrement from maximum remission/response levels in granulocytes or platelets; Reduction in Hgb concentration by ≥ 2 g/dL; Transfusion dependence. Based on Kaplan-Meier Estimates.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 3 | 8 | 7 | 7 | 7 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Months | 1.56 [0.82 to 2.30] | 2.02 [1.94 to 2.10] | 3.99 [0.89 to 7.10] | 0.95 [0.30 to 1.74] | 1.32 [0.79 to 2.79] | 1.02 [0.66 to 5.00] | 1.45 [0.39 to 2.33] | 1.32 [0.30 to 7.10] | 3.39 [0.89 to 3.72] | 1.07 [0.43 to 10.32] | 1.94 [0.95 to 2.33] | 1.51 [0.46 to 2.93] | 0.97 [0.30 to 2.50] | 7.81 [7.59 to 8.02] | 0.99 [0.30 to 2.20] | 0.99 [0.30 to 2.20] | 1.84 [NA to NA] — insufficient number of participants with events

21. Secondary Outcome: Duration of Remission/Response (DOR)
Description: DOR is defined as the time from first remission/response observed to the date of relapse, death or PD. PD=At least 50% decrement from maximum remission/response levels in granulocytes or platelets; Reduction in Hgb concentration by ≥ 2 g/dL; Transfusion dependence. Based on Kaplan-Meier Estimates.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants with response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 8 | 7 | 7 | 9 | 3 | 7 | 8 | 2 | 9 | 9 | 1
Months | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 1.32 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [3.16 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 3.02 [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

22. Secondary Outcome: Time to Remission/Response (TTR)
Description: TTR is defined as the time between the date of first dose and the earliest date any remission/response (any complete remissions or partial remissions or better) is observed. CR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; CRi=residual neutropenia < 1,000 μL, thrombocytopenia < 100,000/μL. CRh=neutrophils ≥ 500μL, platelets ≥500,000μL, blasts <5%; CRc=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; cytogenetics normal; CRm=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%, negative EMD; PR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts decrease in ≥ 50 resulting in 5 to 25%. Based on Kaplan-Meier Estimates.
Time Frame: Up to approximately 25 months after the last dose
Population: All treated participants with available TTR results
Measure: Median (Full Range); unit: Months
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4 | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Months |  |  |  |  | 0.85 [0.85 to 0.85] | 2.01 [2.01 to 2.01] | 1.00 [0.8 to 1.2] |  | 1.12 [0.9 to 1.4] | 1.02 [1.0 to 1.1] |  |  | 1.55 [0.9 to 2.2] |  |  | 0.95 [0.95 to 0.95] |

23. Secondary Outcome: Complete Remission Rate (CRR)
Description: The complete remission rate (CRR) is defined as the percent of participants whose best overall response is any type of Morphologic Complete Remission [CR] (CR, Morphologic Complete Remission with Incomplete Blood Count Recovery (CRi), Morphologic Complete Remission with Partial Hematologic Recovery (CRh), Cytogenetic Complete Remission (CRc) and Molecular Complete Remission (CRm)). CR=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; CRi=residual neutropenia < 1,000/μL, thrombocytopenia < 100,000/μL. CRh=neutrophils ≥ 500μL, platelets ≥500,000μL, blasts <5%; CRc=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%; cytogenetics normal; CRm=neutrophils ≥ 1,000μL, platelets ≥100,000μL, blasts <5%, negative EMD.
Time Frame: Up to approximately 88 months
Population: All treated participants with available CRR results
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 8 | 0 | 0 | 1 | 0
Percent of participants |  |  |  |  | 6.7 [0.17 to 31.95] | 33.3 [0.84 to 90.57] | 25.0 [3.19 to 65.09] |  | 28.6 [3.67 to 70.96] | 22.2 [2.81 to 60.01] |  |  | 12.5 [0.32 to 52.65] |  |  | 11.1 [0.28 to 48.25] |

24. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Transformation
Description: Time to acute AML transformation in part B Myelodysplastic Syndromes (MDS) participants only. Based on Kaplan-Meier Estimates.
Time Frame: Up to approximately 88 months
Population: All treated participants in part B - MDS only as pre-specified
Measure: Median (Full Range); unit: Months
Arm/Group | Part B - MDS 3.6 mg + DEX | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 0
Months | 4.88 [4.6 to 5.1] |

25. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data
Time Frame: Cycle 1 Day 1(C1D1), C1D5, C1D7, C1D8, C1D10,
Population: All treated participants with pharmacokinetic measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 7 | 7 | 7 | 8 | 3 | 7 | 7 | 2 | 8 | 8 | 1
ng/mL
  C1D1: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 7 | 7 | 7 | 8 | 3 | 7 | 7 | 2 | 8 | 7 | 1
  C1D1 | 17.21 (47.65) | 59.61 (19.21) | 71.30 (0.60) | 143.42 (356.59) | 106.23 (88.56) | 94.31 (75.89) | 90.77 (46.38) | 103.00 (26.22) | 122.02 (52.39) | 116.60 (276.56) | 129.53 (61.68) | 96.78 (42.25) | 179.97 (211.30) | 499.18 (2403.37) | 50.99 (59.25) | 73.94 (72.41) | 24.50 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D5: number analyzed (Participants) | 2 | 2 | 2 | 3 | 11 | 1 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D5 | 21.15 (1.67) | 47.19 (55.57) | 33.31 (90.26) | 120.48 (42.56) | 115.40 (93.25) | 82.40 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 147.16 (95.76) | 107.68 (17.50) |  |  |  |  |  |  |  |  |
  C1D7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 1
  C1D7 |  |  |  |  |  |  |  |  | 156.65 (48.38) |  |  |  |  |  | 47.33 (75.83) | 99.57 (79.67) | 108.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D10 |  |  |  |  |  |  |  |  |  | 107.89 (28.36) |  |  |  |  |  |  |
  C1D8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0
  C1D8 |  |  |  |  |  |  |  |  |  |  | 215.18 (17.41) | 111.52 (29.72) |  |  |  |  |

26. Secondary Outcome: Time to Peak Plasma Concentration (Tmax)
Description: Time to peak plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: Cycle 1 Day 1(C1D1), C1D5, C1D7, C1D8, C1D10. 1 cycle = 28 days
Population: All treated participants with pharmacokinetic measurements
Measure: Median (Full Range); unit: hour
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 7 | 7 | 7 | 8 | 3 | 7 | 7 | 2 | 8 | 8 | 1
hour
  C1D1: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 7 | 7 | 7 | 8 | 3 | 7 | 7 | 2 | 8 | 7 | 1
  C1D1 | 0.050 [0.05 to 0.05] | 0.058 [0.05 to 0.07] | 0.042 [0.03 to 0.05] | 0.667 [0.57 to 1.13] | 0.617 [0.25 to 0.98] | 0.250 [0.25 to 0.43] | 0.350 [0.25 to 1.10] | 0.767 [0.67 to 1.33] | 0.750 [0.25 to 0.82] | 0.750 [0.25 to 0.78] | 0.750 [0.25 to 0.75] | 0.783 [0.25 to 0.98] | 0.767 [0.25 to 1.00] | 0.783 [0.77 to 0.80] | 0.783 [0.23 to 1.03] | 0.800 [0.37 to 24.10] | 1.083 [1.083 to 1.083]
  C1D5: number analyzed (Participants) | 2 | 2 | 2 | 3 | 11 | 1 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D5 | 0.050 [0.03 to 0.07] | 0.058 [0.05 to 0.07] | 0.158 [0.05 to 0.27] | 0.783 [0.43 to 0.98] | 0.550 [0.23 to 1.32] | 1.483 [1.483 to 1.483] | 0.383 [0.25 to 2.58] | 0.750 [0.73 to 0.75] |  |  |  |  |  |  |  |  |
  C1D7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 1
  C1D7 |  |  |  |  |  |  |  |  | 0.583 [0.25 to 0.80] |  |  |  |  |  | 1.067 [0.77 to 4.42] | 0.775 [0.60 to 1.12] | 0.667 [0.667 to 0.667]
  C1D10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D10 |  |  |  |  |  |  |  |  |  | 0.800 [0.75 to 1.53] |  |  |  |  |  |  |
  C1D8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0
  C1D8 |  |  |  |  |  |  |  |  |  |  | 0.750 [0.50 to 0.78] | 0.733 [0.28 to 1.00] |  |  |  |  |

27. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Post-dose (AUC 0 - 24)
Description: Area under the plasma concentration-time curve from Time 0 to 24 hours post-dose.
Time Frame: Cycle 1 Day 1(C1D1), C1D5, C1D7, C1D8, C1D10. 1 cycle = 28 days
Population: All treated participants with pharmacokinetic measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 7 | 7 | 7 | 8 | 3 | 7 | 7 | 2 | 8 | 8 | 1
h*ng/mL
  C1D1: number analyzed (Participants) | 2 | 2 | 2 | 7 | 15 | 3 | 7 | 7 | 7 | 8 | 3 | 7 | 7 | 2 | 8 | 7 | 1
  C1D1 | 22.93 (33.59) | 110.11 (68.80) | 121.06 (111.97) | 323.10 (75.44) | 382.59 (37.60) | 486.47 (70.83) | 333.79 (25.04) | 723.89 (30.43) | 618.99 (64.81) | 371.58 (87.80) | 304.37 (43.55) | 487.14 (69.15) | 835.2 (66.9) | 790.5 (250.4) | 245.53 (67.51) | 270.49 (102.71) | 188.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D5: number analyzed (Participants) | 2 | 2 | 2 | 3 | 10 | 1 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D5 | 26.94 (35.62) | 141.84 (99.49) | 142.54 (148.76) | 769.03 (25.72) | 536.30 (39.55) | 1360.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 624.30 (55.31) | 669.55 (23.92) |  |  |  |  |  |  |  |  |
  C1D7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 1
  C1D7 |  |  |  |  |  |  |  |  | 959.76 (80.24) |  |  |  |  |  | 369.61 (48.65) | 409.43 (54.13) | 425.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D10 |  |  |  |  |  |  |  |  |  | 777.69 (14.64) |  |  |  |  |  |  |
  C1D8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0
  C1D8 |  |  |  |  |  |  |  |  |  |  | 422.26 (41.02) | 648.01 (35.29) |  |  |  |  |

28. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2)
Description: Terminal phase elimination half-life calculated as [(ln 2)/λz], where λz is the apparent terminal rate constant. t1/2 will only be calculated when a reliable estimate for λz can be obtained.
Time Frame: Cycle 1 Day 1(C1D1) and C1D5. 1 cycle = 28 days
Population: All treated participants with pharmacokinetic measurements
Measure: Median (Full Range); unit: hour
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 2 | 6 | 6 | 7 | 8 | 3 | 7 | 7 | 2 | 6 | 6 | 1
hour
  C1D1 | 3.783 [2.61 to 4.96] | 7.717 [6.43 to 9.01] | 7.295 [3.60 to 10.99] | 5.991 [3.92 to 11.88] | 6.317 [3.68 to 10.61] | 6.864 [4.97 to 8.76] | 4.001 [3.70 to 4.98] | 8.378 [5.35 to 13.45] | 6.584 [3.86 to 8.54] | 3.739 [3.46 to 11.48] | 4.649 [4.28 to 5.61] | 6.795 [3.51 to 9.75] | 6.246 [3.01 to 15.47] | 6.844 [4.74 to 8.94] | 6.432 [2.47 to 8.39] | 4.800 [3.50 to 10.78] | 7.737 [7.737 to 7.737]
  C1D5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Total Body Clearance (CL)
Description: Total plasma clearance after IV administration, calculated as [Dose/ AUC(INF)] following single administration, and [Dose/ AUC(0-24)] at steady state.
Time Frame: Cycle 1 Day 1(C1D1), C1D5, C1D7, C1D8, C1D10. 1 cycle = 28 days
Population: All treated participants with pharmacokinetic measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 2 | 7 | 6 | 7 | 8 | 3 | 7 | 7 | 2 | 6 | 8 | 1
L/h
  C1D1: number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 2 | 6 | 6 | 7 | 8 | 3 | 7 | 7 | 2 | 6 | 6 | 1
  C1D1 | 12.684 (38.525) | 4.868 (75.331) | 8.796 (143.853) | 6.882 (74.110) | 7.352 (43.454) | 6.140 (125.199) | 11.105 (24.102) | 5.932 (24.699) | 5.418 (69.589) | 7.551 (94.257) | 9.618 (42.482) | 6.828 (77.163) | 3.809 (71.852) | 4.359 (265.439) | 9.817 (73.556) | 11.494 (105.754) | 9.350 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D5: number analyzed (Participants) | 2 | 2 | 2 | 3 | 10 | 1 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D5 | 11.134 (35.442) | 4.238 (99.224) | 8.423 (149.082) | 3.120 (25.689) | 5.594 (39.561) | 2.650 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 5.772 (55.283) | 6.721 (23.895) |  |  |  |  |  |  |  |  |
  C1D7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 8 | 1
  C1D7 |  |  |  |  |  |  |  |  | 3.751 (80.086) |  |  |  |  |  | 5.910 (44.624) | 6.615 (57.381) | 7.060 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C1D10 |  |  |  |  |  |  |  |  |  | 3.857 (14.571) |  |  |  |  |  |  |
  C1D8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0
  C1D8 |  |  |  |  |  |  |  |  |  |  | 7.098 (40.903) | 5.553 (35.415) |  |  |  |  |

30. Secondary Outcome: Volume of Distribution (Vz)
Description: Volume of distribution calculated at first dose only. Calculated as [Vz = Dose/ AUC(INF) * λz for Day 1].
Time Frame: Cycle 1 Day 1(C1D1) and C1D5. 1 cycle = 28 days
Population: All treated participants with pharmacokinetic measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 14 | 2 | 6 | 6 | 7 | 8 | 3 | 7 | 7 | 2 | 6 | 6 | 1
L
  C1D1 | 65.74 (8.29) | 53.38 (45.41) | 79.87 (27.70) | 64.51 (82.15) | 68.28 (32.16) | 58.48 (62.34) | 65.80 (20.59) | 70.30 (28.14) | 46.58 (41.72) | 55.03 (73.60) | 66.95 (55.61) | 60.12 (41.69) | 33.559 (70.261) | 40.973 (129.680) | 77.996 (37.418) | 86.419 (99.105) | 104.000 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  C1D5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Renal Clearance (CLr)
Description: Renal clearance of CC-90009 (CLr)
Time Frame: Cycle 1 Day 1(C1D1). 1 cycle = 28 days
Population: All treated participants with pharmacokinetic measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part A - 0.3 mg | Part A - 0.6 mg | Part A - 1.2 mg | Part A - 2.4 mg | Part A - 3.0 mg | Part A - 3.6 mg | Part A - 3.6 mg + DEX | Part A - 4.5 mg | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - AML 3.6 mg + DEX | Part B - MDS 3.6 mg + DEX | Part B - AML 2.4 mg | Part B - AML 3.0 mg | Part B - MDS 3.0 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 2 | 6 | 6 | 1
L/h |  |  |  |  | 0.63900 (200.50356) |  |  |  |  |  | 0.61571 (219.79379) | 1.10066 (38.74255) |  | 40.973 (129.680) | 77.996 (37.418) | 86.419 (99.105) | 104.000 (NA) — Insufficient number of participants to calculate geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 76 months). SAEs and Other AEs were assessed from first dose to 28 days post the last dose (up to approximately 25 months).
Groups:
- Part A - 0.3 mg (Days 1 - 5 of 28): Part A - CC-90009 QD 0.3 mg (Days 1 - 5 of 28)
- Part A - 0.6 mg (Days 1 - 5 of 28): Part A - CC-90009 QD 0.6 mg (Days 1 - 5 of 28)
- Part A - 1.2 mg (Days 1 - 5 of 28): Part A - CC-90009 QD 1.2 mg (Days 1 - 5 of 28)
- Part A - 2.4 mg (Days 1 - 5 of 28): Part A - CC-90009 2.4 mg (Days 1 - 5 of 28)
- Part A - 3.0 mg (Days 1 - 5 of 28): Part A - CC-90009 QD 3.0 mg (Days 1 - 5 of 28)
- Part A - 3.6 mg (Days 1 - 5 of 28): Part A - CC-90009 QD 3.6 mg (Days 1 - 5 of 28)
- Part A - 3.6 mg + DEX (Days 1 - 5 of 28): Part A - CC-90009 QD 3.6 mg + Dexamethasone 10 mg IV (Days 1 - 5 of 28)
- Part A - 4.5 mg (Days 1 - 5 of 28): Part A - CC-90009 daily (QD) 4.5 mg (Days 1 - 5 of 28)
- Part B - 3.6 mg + DEX (Days 1 - 5 of 28); Part B - MDS 3.6 mg + DEX (Days 1 - 5 of 28): Part B - MDS CC-90009 3.6 mg + Dexamethasone (Days 1 - 5 of 28)
- Part B - 2.4 mg (Days 1 - 7 of 28): Part B - MDS CC-90009 24 mg (Days 1 - 7 of 28)
- Part B - 3.0 mg (Days 1 - 7 of 28): Part B - CC-90009 3.0 mg (Days 1 - 7 of 28)
- Part B - MDS 3.0 mg (Days 1 - 7 of 28): Part B - MDS CC-90009 3.0 mg (Days 1 - 7 of 28)
Arm/Group | Part A - 0.3 mg (Days 1 - 5 of 28) | Part A - 0.6 mg (Days 1 - 5 of 28) | Part A - 1.2 mg (Days 1 - 5 of 28) | Part A - 2.4 mg (Days 1 - 5 of 28) | Part A - 3.0 mg (Days 1 - 5 of 28) | Part A - 3.6 mg (Days 1 - 5 of 28) | Part A - 3.6 mg + DEX (Days 1 - 5 of 28) | Part A - 4.5 mg (Days 1 - 5 of 28) | Part A - 3.6 mg (Days 1 - 7 of 28) | Part A - 3.0 mg (Days 1- 10 of 28) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) | Part B - 3.6 mg + DEX (Days 1 - 5 of 28) | Part B - MDS 3.6 mg + DEX (Days 1 - 5 of 28) | Part B - 2.4 mg (Days 1 - 7 of 28) | Part B - 3.0 mg (Days 1 - 7 of 28) | Part B - MDS 3.0 mg (Days 1 - 7 of 28)
All-Cause Mortality (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 7/7 | 14/15 | 2/3 | 8/8 | 6/7 | 7/7 | 7/9 | 2/3 | 7/7 | 8/8 | 2/2 | 9/9 | 9/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 1/2 | 6/7 | 15/15 | 3/3 | 7/8 | 7/7 | 7/7 | 6/9 | 3/3 | 6/7 | 8/8 | 1/2 | 9/9 | 8/9 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 7/7 | 15/15 | 3/3 | 8/8 | 7/7 | 7/7 | 9/9 | 3/3 | 7/7 | 8/8 | 2/2 | 8/9 | 9/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - 0.3 mg (Days 1 - 5 of 28) (N=2) | Part A - 0.6 mg (Days 1 - 5 of 28) (N=2) | Part A - 1.2 mg (Days 1 - 5 of 28) (N=2) | Part A - 2.4 mg (Days 1 - 5 of 28) (N=7) | Part A - 3.0 mg (Days 1 - 5 of 28) (N=15) | Part A - 3.6 mg (Days 1 - 5 of 28) (N=3) | Part A - 3.6 mg + DEX (Days 1 - 5 of 28) (N=8) | Part A - 4.5 mg (Days 1 - 5 of 28) (N=7) | Part A - 3.6 mg (Days 1 - 7 of 28) (N=7) | Part A - 3.0 mg (Days 1- 10 of 28) (N=9) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) (N=3) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) (N=7) | Part B - 3.6 mg + DEX (Days 1 - 5 of 28) (N=8) | Part B - MDS 3.6 mg + DEX (Days 1 - 5 of 28) (N=2) | Part B - 2.4 mg (Days 1 - 7 of 28) (N=9) | Part B - 3.0 mg (Days 1 - 7 of 28) (N=9) | Part B - MDS 3.0 mg (Days 1 - 7 of 28) (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 5 | 2 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Citrobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stenotrophomonas sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 3 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - 0.3 mg (Days 1 - 5 of 28) (N=2) | Part A - 0.6 mg (Days 1 - 5 of 28) (N=2) | Part A - 1.2 mg (Days 1 - 5 of 28) (N=2) | Part A - 2.4 mg (Days 1 - 5 of 28) (N=7) | Part A - 3.0 mg (Days 1 - 5 of 28) (N=15) | Part A - 3.6 mg (Days 1 - 5 of 28) (N=3) | Part A - 3.6 mg + DEX (Days 1 - 5 of 28) (N=8) | Part A - 4.5 mg (Days 1 - 5 of 28) (N=7) | Part A - 3.6 mg (Days 1 - 7 of 28) (N=7) | Part A - 3.0 mg (Days 1- 10 of 28) (N=9) | Part A - 3.0 mg (Day 1 - 3 & Day 8 - 10 of 28) (N=3) | Part A - 3.6 mg (Day 1 - 3 & Day 8 - 10 of 28) (N=7) | Part B - 3.6 mg + DEX (Days 1 - 5 of 28) (N=8) | Part B - MDS 3.6 mg + DEX (Days 1 - 5 of 28) (N=2) | Part B - 2.4 mg (Days 1 - 7 of 28) (N=9) | Part B - 3.0 mg (Days 1 - 7 of 28) (N=9) | Part B - MDS 3.0 mg (Days 1 - 7 of 28) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 3 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dilated cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 4 | 1 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 10 | 3 | 5 | 6 | 7 | 4 | 2 | 2 | 3 | 2 | 5 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 5 | 9 | 1 | 4 | 6 | 5 | 6 | 3 | 4 | 3 | 2 | 4 | 7 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 8 | 1 | 2 | 2 | 4 | 4 | 2 | 3 | 1 | 0 | 3 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 4 | 4 | 2 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 5 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 3 | 0
Pain (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 4 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Gallbladder oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine storm (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 4 | 2 | 1 | 0 | 4 | 0 | 0 | 4 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 3 | 1 | 4 | 4 | 2 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 2 | 1 | 5 | 3 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood parathyroid hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calcium ionised decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coagulation time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Electrocardiogram QT shortened (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 4 | 1 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 2 | 2 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 5 | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 5 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 11 | 3 | 6 | 7 | 7 | 8 | 3 | 5 | 6 | 2 | 5 | 7 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 3 | 2 | 3 | 2 | 5 | 1 | 0 | 4 | 4 | 1 | 1 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 3 | 2 | 2 | 2 | 2 | 3 | 0 | 3 | 3 | 0 | 3 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 4 | 1 | 0 | 1 | 3 | 3 | 0 | 4 | 2 | 1 | 2 | 2 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Refeeding syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 2 | 3 | 0 | 1 | 2 | 1 | 1 | 4 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 2 | 3 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 9 | 2 | 4 | 6 | 6 | 5 | 0 | 1 | 4 | 1 | 2 | 3 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT02848001/Prot_SAP_000.pdf